CLINICAL TRIAL: NCT06624332
Title: Digital Screening and Brief Intervention for Perinatal Substance Use in Home Visiting
Brief Title: Home Visitation Enhancing Linkages Project in Kansas
Acronym: HELP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Sarah Dauber, Vice President, The National Center on Addiction and Substance Abuse at Columbia University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HELP 3.0 Kansas; R34DA061238 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No intervention Routine HV Only (No Intervention): Routine home visiting only
- e-SBI main session (Experimental): e-SBI main session
  Interventions: Behavioral: e-SBI main session
- e-SBI main session + booster (Experimental): e-SBI main session and e-SBI booster session
  Interventions: Behavioral: e-SBI main session; Behavioral: e-SBI Booster Session
- Text messaging only (Experimental): text messaging
  Interventions: Behavioral: Text messaging
- e-SBI main session + text messaging (Experimental): e-SBI main session Text messaging
  Interventions: Behavioral: e-SBI main session; Behavioral: Text messaging
- e-SBI main + e-SBI booster + text messaging (Experimental): e-SBI main session e-SBI booster session text messaging
  Interventions: Behavioral: e-SBI main session; Behavioral: e-SBI Booster Session; Behavioral: Text messaging

INTERVENTIONS:
Behavioral: e-SBI main session — Single 20-minute e-SBI session that includes screening followed by brief motivational intervention.
  Arms: e-SBI main + e-SBI booster + text messaging; e-SBI main session; e-SBI main session + booster; e-SBI main session + text messaging
Behavioral: e-SBI Booster Session — A 20-minute booster e-SBI session that reinforces content from the main e-SBI session.
  Arms: e-SBI main + e-SBI booster + text messaging; e-SBI main session + booster
Behavioral: Text messaging — 4 weeks of daily automated text messages that reinforce content from the e-SBI main session.
  Arms: Text messaging only; e-SBI main + e-SBI booster + text messaging; e-SBI main session + text messaging

SUMMARY:
The goal of this study is to learn about whether digital screening and brief intervention can help address substance use in postpartum mothers who are enrolled in home visiting programs. The main questions it aims to answer are:

1. What combination of digital intervention components work best for postpartum mothers in home visiting programs?
2. What are the factors that help the intervention work best in home visiting, and what factors serve as barriers to the success of the intervention? Participants in the study will include home visiting staff and postpartum home visiting clients.

Participants who are home visitors will be asked to participate in focus groups and interviews, introduce the study to their clients and refer interested clients to the study, complete online surveys, and implement the home visitor components of the intervention with their clients who enroll in the study.

Participants who are home visiting clients will be asked to participate in focus groups and interviews, complete online surveys, and complete the digital screening and brief intervention sessions.

DETAILED DESCRIPTION:
The postpartum period is a time of significant risk for substance use (SU), as more than half of women who reduce their SU during pregnancy return to pre-pregnancy levels within 3 months postpartum, due to hormonal changes, the stress of caring for a newborn, sleep deprivation, and social isolation1,2. Postpartum SU may increase risk for child maltreatment, which can have devastating impacts on brain development, leading to long-term impairment3-6,7. Effective treatments for SU exist, but are often not accessed by postpartum mothers due to stigma and fear of child removal8. Brief interventions delivered during the early postpartum period may prevent postpartum escalation of SU, but often do not reach those at highest risk, and when they do, effects are short-lived9,10. There is a critical need to determine the most effective approaches for reaching high-risk new mothers to provide evidence-based interventions to prevent postpartum SU.

Home visiting (HV), a strategy for delivering voluntary preventive services aimed at optimizing parent and child outcomes across the life course, is the primary supportive intervention offered to at-risk families during the perinatal period in the United States11,12. As HV is often one of the only service touchpoints for vulnerable families during the postpartum period, it is a promising venue for reaching new mothers to prevent risks associated with SU. However, the most widely used HV models do not have standardized protocols for identifying and addressing SU risk, beyond making referrals to community based services13, which leaves many mothers with unaddressed SU concerns that put themselves and their babies at risk. Our team has been working to fill this significant gap in services since 2013, and this study represents the next phase of our work, ultimately aimed at providing the HV field with a feasible and effective tool for managing perinatal SU and reducing associated risks to families.

Screening, Brief Intervention, and Referral to Treatment (SBIRT), originally designed to reduce gaps in the service continuum from primary care to SU treatment14,15, has been widely recommended as a public health model for addressing SU16-19. This approach may be a good fit for the HV context given its non-judgmental nature, the prevalence of low-to-moderate risk among HV clients, and the small proportion of HV clients who are actively seeking SU treatment20,21. Two key challenges preclude the successful integration of traditional SBIRT procedures into HV. First, HV clients are often reluctant to disclose SU to professionals, including HVrs, due to shame, stigma, denial, and fear of child removal22-25. Second, most HVrs are lay professionals, who lack the advanced clinical training and skills needed to effectively deliver evidence-based brief interventions (BI)26.

Screening and Brief Intervention (SBI) that is delivered digitally via computer or smartphone has great potential to overcome both of these challenges, as it does not require clients to directly disclose SU to a provider or providers to deliver evidence-based BIs. Digital SBI has been proven accessible and highly acceptable in postpartum mothers when delivered in healthcare settings, but shows small and inconsistent effects27,28. The BI literature suggests that extended intervention contacts may bolster BI effects29,30. Additional digital BI sessions and automated text messages are potential methods of extending BI impacts, and both have demonstrated acceptability in postpartum mothers. In a prior study, we developed an innovative digital SBI model that was tailored to the HV context (SBI-HV) that included an electronic SBI (e-SBI) that clients completed on their smartphones in between home visits, and a home visitor facilitation component to promote integration of the e-SBI into routine HV. The e-SBI applied motivational interviewing (MI) principles and the Feedback, Responsibility, Advice, Menu Options, Empathy, and Self-Efficacy BI framework. Confidentiality and preserving clients' choice regarding disclosing SU to their home visitor is core to SBI-HV. A small pilot study supported initial feasibility and acceptability of SBI-HV. Building on our prior R34, the proposed study aims to further optimize the SBI-HV by applying a factorial design to compare preliminary impacts of three SBI-HV delivery strategies: a single e-SBI session (main e-SBI), the main e-SBI session plus a booster session (booster e-SBI), and 4 weeks of tailored text messaging following e-SBI (text messaging). Additionally, we will systematically assess implementation facilitators and barriers to inform development of targeted implementation strategies to support sustainable integration of SBI-HV into routine HV.

The proposed R34 will use a Type 1 hybrid implementation-effectiveness design with a pilot 3X2 factorial trial and apply the RE-AIM and PRISM implementation frameworks to achieve the following specific aims:

1. Test the impact of 3 SBI-HV delivery strategies (main e-SBI; main e-SBI + booster e-SBI; and text messaging) on postpartum SU, maternal self-efficacy, motivation to avoid SU, and HV retention.
2. Evaluate feasibility, acceptability, fidelity, and facilitators and barriers to the 3 SBI-HV delivery strategies.
3. Develop tailored implementation strategies to support SBI-HV integration into routine HV.

We will partner with the Kansas Healthy Families (HF) multi-site HV system to complete study aims in 3 phases. All phases will be guided by the RE-AIM and PRISM implementation frameworks.

Phase 1: Pre-Implementation (Months 1-6): We will conduct a mixed-methods assessment of PRISM domains to inform SBI-HV implementation. Participants will include 36 home visitors, 36 clients, 12 supervisors, and 12 administrative staff representing all 12 Kansas HF programs. During this phase, we will assess program capacity and readiness to implement SBI-HV with the following goals: (a) select implementation program sites; (b) promote buy-in from key program staff; and (c) inform local adaptations to the SBI-HV.

Phase 2: Implementation (Months 7-25): We will conduct a pilot 3X2 factorial trial with 120 clients and 20 home visitors at 5 sites to obtain proof-of-concept data on the individual and combined impacts of the SBI-HV delivery strategies (main e-SBI, main e-SBI + booster, and text messaging) on SU, motivation, self-efficacy, and HV retention, as well as quantitative data on the RE-AIM domains.

Phase 3: Post-Implementation (Months 26-36): We will conduct qualitative interviews with home visitors, clients, supervisors, and administrative staff who participated in the factorial trial to systematically assess implementation facilitators and barriers using the RE-AIM and PRISM frameworks. Following assessment, we will conduct an iterative stakeholder-engaged process of developing candidate implementation strategies for testing in a future study.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age 18 years old or older
* Gave birth to a baby within the prior year
* Enrolled in a Healthy Families Kansas program with a participating home visitor
* Not currently enrolled in substance use treatment

Exclusion Criteria:

* Does not speak English
* Under age 18 years
* Did not give birth to a baby within the prior year
* Not enrolled in a Healthy Families Kansas program with a participating home visitor
* Currently enrolled in substance use treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In order to be eligible, participants must have given birth to a baby in the prior year. Thus, their biological sex must be female, but biological females who express their gender identity in other ways are still eligible, as long as they gave birth to a baby in the prior year.
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Substance use | Assessed at 3-month follow-up and 6-month follow-up
  Quantity and frequency of substance use, measured by the Timeline Follow Back.

SECONDARY OUTCOMES:
Motivation to avoid substance use | Assessed at 3-month follow-up and 6-month follow-up
  How motivated are you to avoid substance use until your baby is one year old, on a scale of 1 to 10. This Maternal Motivation Scale was developed by Ondersma and has been widely used in studies of brief digital interventions for perinatal substance use.
Maternal self-efficacy | Assessed at 3-month and 6-month follow-up
  Confidence in your ability to care for your baby, assessed via the Karitane Parenting Confidence Scale.
Home visiting retention | Assessed at 6-month follow-up
  Length of time enrolled in the home visiting program in months.